

Official Title: Oxygen Reserve Index Validation

for RD Lite Sensors

Date of Statistical Plan: August 1, 2017

NCT Number: NCT03128892

## **Statistical Analysis Plan**

Specificity, Sensitivity and Concordance were used as metrics for evaluation. They are computed using the following formulas:

Specificity = N1/(N1 + N4)

Sensitivity = N3 / (N2 + N3)

Concordance = (N1 + N3) / (N1 + N2 + N3 + N4)

where N1, N2, N3 and N4 are defined as per the figure below



 $\Delta PaO_2$  and  $\Delta ORI$  are defined as shown below:

$$\Delta PaO_2 = PaO_2(t) - PaO_2(t_{ref})$$

$$\Delta ORI = ORI(t) - ORI(t_{ref})$$